CLINICAL TRIAL: NCT02888041
Title: Is There an Interest in Repeating the Vaginal Administration of Dinoprostone (Propess®), to Promote Induction of Labor of Pregnant Women at Term?
Acronym: RE-DINO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not enough patients
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I15014 (RE-DINO)
Record Dates: First submitted 2016-08-24; First posted 2016-09-02 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Cervical Ripening; Pregnancy
Keywords: Cervical ripening; Pregnancy; Vaginal Administration
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dinoprostone (Experimental): In case of failure of cervical ripening after a first intravaginal delivery device of Dinoprostone (Propess® 10 mg), patients receive a second Propess®, followed by Oxytocin 5U.I/ml (Syntocinon®) (if necessary) and epidural analgesia if desired by the patient.
  Interventions: Drug: Dinoprostone
- Oxytocine (Active Comparator): In case of failure of cervical ripening after a first intravaginal delivery device of Dinoprostone (Propess® 10mg), patients receive directly Oxytocin 5U.I/ml (Syntocinon®) and epidural analgesia if desired by the patient.
  Interventions: Drug: Oxytocine

INTERVENTIONS:
Drug: Dinoprostone — In case of failure of cervical ripening after a first intravaginal delivery device of Dinoprostone (Propess® 10 mg), patients receive a second Propess®, followed by Oxytocin 5U.I/ml (Syntocinon®) (if necessary) and epidural analgesia if desired by the patient.
  Arms: Dinoprostone
Drug: Oxytocine — In case of failure of cervical ripening after a first intravaginal delivery device of Dinoprostone (Propess® 10mg), patients receive directly Oxytocin 5U.I/ml (Syntocinon®) and epidural analgesia if desired by the patient.
  Arms: Oxytocine

SUMMARY:
According perinatal surveys, induction of labor is performed at more than 20% of pregnant women.

According to a survey on the trigger practices in France, prostaglandins are widely used to initiate cervical ripening, usually by laying intravaginal dinoprostone (Propess®).

The overall work-up rate due to the use of a single Propess® is 74.6% with 80% of vaginal deliveries.

Currently, 25.4% of patients who was not put in work after 24 hours are triggered by oxytocin (Syntocinon®) or directly caesarean. The initial installation of intravaginal dinoprostone limits the use of oxytocin (Syntocinon®) or in lower doses.

Using a second Propess® is carried out in several maternity hospitals, as reported by the survey on the cervical ripening practices in France. This second administration could be the solution to reduce the rate of caesarean in France which amounted to 20.8%.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is >=18 years.
* Term pregnancy > 37 weeks
* Induction of labor in progress, medically indicated
* Patients who have had the establishment of a first Propess®, within 24 to 36 hours (before signing the consent)
* Cephalic presentation
* Unfavorable cervical conditions (Bishop score <6) 1 hour prior to inclusion
* Intact Membranes
* Affiliated with a social security system
* Having signed the consent form.

Exclusion Criteria:

* Multiple pregnancy
* Uterus scar
* Contraindications to epidural anesthesia
* Contraindications to Propess®: recent history of pelvic inflammatory disease; hypersensitivity to prostaglandins Adverse effects appeared in the first Propess®: anaphylactic shock, disseminated intravascular coagulation (DIC).
* Contraindications to Syntocinon: Hypersensitivity to oxytocin, cardiovascular disorders and severe toxemia of pregnancy.
* Contraindications to vaginal delivery (placenta previa, previa obstacle ...)
* Premature Rupture of Membranes (PROM)
* Intra Uterine Growth Retardation (IUGR) <3rd percentile
* Macrosomia> 97th percentile
* Severe Impaired fetal heart rate
* In Utero Fetal Death (IUFD)
* Medical Termination of pregnancy or lethal fetal pathology
* Patient under guardianship or trusteeship safeguard justice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-04-23 (Actual); Study Completion 2022-04-23 (Actual)

PRIMARY OUTCOMES:
Rate of deliveries vaginally | At delivery
  The rate of births vaginally in each arm

SECONDARY OUTCOMES:
Failure of induction of labor | At delivery
  The failure of induction of labor correspond to cervical dilation remaining <3cm despite 6 hours of Syntocinon (or 1 syringe) and regular uterine contractions and amniotomy.
  The success of the trigger is defined by regular uterine contractions and cervical dilatation ≥ 3 cm.
Time of work | delivery time
  Time in minutes between the start of work defined by the onset of regular uterine contractions and cervical dilation ≥3 cm and delivery.
Caesarean indications | At delivery
  Caesarean indications
Proportion of instrumental delivery | At delivery
  The proportion of instrumental delivery
Proportion of complications of delivery and various care. | Day 1
  The proportion of complications of delivery and various care.
Proportion of complete uterine rupture | At delivery
  The proportion of complete uterine rupture
Transfer in Intensive Care Unit | 10 Days
  The transfer in Intensive Care Unit
Maternal death | 10 Days
  Maternal death
Hospital stay of mother | 10 Days
  Hospital stay of mother
Apgar score | 3 Min, 5 Min and 10 Min
  Determination of Apgar score
Visual estimation of presence of amniotic fluid meconium | At the birth
  Visual estimation of presence of meconium in amniotic fluid. Absence of meconium if transparent and presence if colored.
Proportion of transfer neonatal or newborn intensive care unit | At the birth
  The proportion of transfer neonatal or newborn intensive care unit
Fetal / neonatal death | At the birth
  Fetal / neonatal death
Assessment of fetal acidosis by measuring of pH, lactates and base excess | At the birth
  Assessment of fetal acidosis by measuring of pH, lactates and base excess

CONTACTS AND LOCATIONS:
Overall Officials: Perrine COSTE-MAZEAU, MD, Principal Investigator — University Hospital, Limoges
Locations (7):
- France (7):
  - CH de Blois, Blois
  - CH de BRIVE, Brive-la-Gaillarde
  - CH Metropole Savoie, Chambéry
  - Hôpital d'Estaing - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de LIMOGES, Limoges
  - Hôpital Nord - APHM, Marseille
  - CH de TULLE, Tulle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coste Mazeau P, Hessas M, Martin R, Eyraud JL, Margueritte F, Aubard Y, Sallee C, Sire F, Gauthier T. Is there an interest in repeating the vaginal administration of dinoprostone (Propess(R)), to promote induction of labor of pregnant women at term? (RE-DINO): study protocol for a randomized controlled trial. Trials. 2020 Jan 8;21(1):51. doi: 10.1186/s13063-019-3985-0. PMID 31915047